CLINICAL TRIAL: NCT06376487
Title: Evaluation of Pulmonary Aeration and Muscle Thickening Fraction in Infants With Bronchiolitis Using a High-flow Nasal Cannula: Association of Electrical Impedance Tomography and Ultrasound
Brief Title: Pulmonary Aeration and Muscle Thickening Fraction: Association of Electrical Impedance Tomography and Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 75202423.2.0000.0071
Record Dates: First submitted 2024-02-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-02

CONDITIONS: Bronchiolitis
Keywords: Pulmonary;; Ventilation;
MeSH Terms: conditions — Bronchiolitis; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: A prospective clinical study to evaluated four different flow rate in infants with bronchiolitis using high flow nasal cannula
Masking Description: Patient will not know the flow rate sequence used during the assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- flow rate sequence (Experimental): Four different randomized flow rates will be used for evaluation: 2.0 liter.Kg-1.min-1, 1.5 liter.Kg-1.min-1, 1.0 liter.Kg-1.min-1, 0.5 liter.Kg-1.min-1. At the end of the randomized order evaluation the infant will remain in the flow of 0.5 liter.Kg-1.min-1 for 5 minutes and then return to the flow of 2.0 liter.Kg-1.min-1. The EIT parameters, ultrasound assessment, and clinical variables will be collected at the end of the 5-minute stay in each lane.
  Interventions: Device: Flow rate evaluation

INTERVENTIONS:
Device: Flow rate evaluation — Four different randomized flow rates will be used for evaluation: 2.0 liter.Kg-1.min-1, 1.5 liter.Kg-1.min-1, 1.0 liter.Kg-1.min-1, 0.5 liter.Kg-1.min-1. At the end of the randomized order evaluation the infant will remain in the flow of 0.5 liter.Kg-1.min-1 for 5 minutes and then return to the flow of 2.0 liter.Kg-1.min-1. The EIT parameters, ultrasound assessment, and clinical variables will be collected at the end of the 5-minute stay in each lane.

SUMMARY:
The goal of this prospective clinical study is to evaluate the effect of different High Flow Nasal Cannula (HFNC) flow rates on diaphragm, rectoabdominal, and oblique thickening fraction, and to determine whether this effect depends on the action of HFNC flow rates on Functional Residual Capacity (FRC) in Infants under 2 years of age with a diagnosis of bronchiolitis and indication for use of HFNC. The main question[s] it aims to answer are:

* If the thickening fraction of the abdominal muscle and diaphragm will change at the different flow rates evaluated
* If the end-expiration lung impedance (EELZ) will change at the different flow rates evaluated

The belt will be installed around the chest before the start of the change in flow rates and monitoring with Electrical Impedance Tomography (EIT) will be initiated. Patients will be positioned in dorsal decubitus elevated 10 to 20 degrees and monitoring will be performed continuously during all flow rate variations and also during the ultrasound performance.

Four different randomized flow rates will be used for evaluation: 2.0 liter.Kg-1.min-1, 1.5 liter.Kg-1.min-1, 1.0 liter.Kg-1.min-1, 0.5 liter.Kg-1.min-1. At the end of the randomized order evaluation the infant will remain in the flow of 0.5 liter.Kg-1.min-1 for 5 minutes and then return to the flow of 2.0 liter.Kg-1.min-1. The EIT parameters, ultrasound assessment, and clinical variables will be collected at the end of the 5-minute stay in each lane.

The randomization of the order of application of the phases will be carried out in blocks, so that the homogeneity of the sequences is maintained even if the collection is interrupted before reaching the total number of individuals. The blocks will be of size two and four and the test and production lists will be generated with the help of the R packages.

DETAILED DESCRIPTION:
OBJECTIVES Main Objective To evaluate, in infants with respiratory failure secondary to bronchiolitis, the effect of different High Flow Nasal Cannula (HFNC) flow rates on diaphragm, rectoabdominal, and oblique thickening fraction, and to determine whether this effect depends on the action of HFNC flow rates on Functional Residual Capacity (FRC).

Secondary Objectives

* To evaluate whether there is a correlation between thickening fraction and respiratory distress score.
* To find values from the EIT data and the thickening fraction that can correlate with possible failure criteria for HFNC therapy.

  5. METHODS 5.1 Study Type and Location A prospective clinical study will be conducted in the Pediatric ICU of Hospital Israelite Albert Einstein from January 2024 to December 2025 5.2 Ethical Aspects This study will be submitted to the Ethics and Research Committee of the Hospital Israelite Albert Einstein. The risk of participating in this research is considered minimal, limited to the accidental loss of confidentiality of the data collected or to skin erythema at the site of application of the belt. Only after signing the informed consent form will the patient be prepared for the beginning of monitoring (Appendix 1) Protocol The tape will be installed around the chest before the start of the change in flow rates and monitoring with EIT will be initiated. Patients will be positioned in dorsal decubitus elevated 10 to 20 degrees and monitoring will be performed continuously during all flow rate variations and also during the ultrasound performance.

Four different randomized flow rates will be used for evaluation: 2.0 liter.Kg-1.min-1, 1.5 liter.Kg-1.min-1, 1.0 liter.Kg-1.min-1, 0.5 liter.Kg-1.min-1. At the end of the randomized order evaluation the infant will remain in the flow of 0.5 liter.Kg-1.min-1 for 5 minutes and then return to the flow of 2.0 liter.Kg-1.min-1. The EIT parameters, ultrasound assessment, and clinical variables will be collected at the end of the 5-minute stay in each lane.

5.5 Randomization: Randomization process The sequence of the flow values will be done using a tool software R 5.6 Clinical and demographic variables Demographic variables such as age, sex, Pediatric Index of Mortality Score (PIM2) (23) and viral screening will be collected when requested during routine hospitalization.

Of the clinical variables, respiratory rate (RR) will be assessed by counting the inspiratory cycles produced by EIT plethysmography in one minute. Heart rate (HR) and peripheral oxygen saturation (SpO2) will be obtained directly from the Infinity Delta multiparameter monitor (Dräger, Lubeck, Germany). Inspired oxygen fraction (FiO2). The Respiratory and Oxygenation Index (ROX index) will also be calculated, which is calculated by the ratio of SpO2/FiO2 by RR.

To evaluate respiratory distress, the investigators will use the respiratory distress score.

Electrical Impedance Tomography The recording of the electrical impedance variation over time is called plethysmogram and this provides information on the ventilation variation which is called Delta Z (∆Z) and has an excellent correlation with the volume variation assessed by computed tomography (25) and the minimum impedance (ZMIN) or ∆EELZ (end-expiration lung impedance) which is the baseline of the plethysmogram and corresponds to the FRC (26,27).

The unit of measurement commonly used to quantify changes in impedance amplitude is arbitrary unit (AU).The average of at least 5 sequential respiratory cycles for each patient, in each flow range, will be considered for evaluation, considering the moment of greatest stability within the final minute of the flow rate to be evaluated. Calculations to obtain delta Z were performed by subtracting the final moment of inspiration from the final moment of expiration. The changes in EELZ (∆EELZ) will be compared to the average EELZ at a flow rate of 0.5 L-kg-1-min-1 (reference flow rate). Therefore, by definition, the average ∆EELZ at the 0.5 L-kg-1-min-1 flow rate will be equal to zero. To obtain clinically meaningful values instead of AU values, the ∆EELZ will be normalized by the corresponding Delta Z at the reference flow rate (28). With this transformation, ∆EELZ can be interpreted as changes in lung aeration measured in multiples of Delta Z (tidal volumes). For example, if an infant has a mean Delta Z of 15 AU at flow rate of 0.5 L-kg-1-min-1, a ∆EELZ of 30 AU at flow rate of 2.0 L-kg-1-min-1 will be shown as 2 (an increase in lung volume twice the Delta Z at the reference flow rate).

Evaluation by ultrasound Serial measurements of thickness and thickening fraction of the diaphragm and abdominal muscle (rectus and oblique) will be collected through ultrasound images by previously trained staff. The images will be taken in the SonoSite M-Turbo® device, using an L25x (13-6 MHz) linear transducer. Heated water-based gel will be used for image acquisition.

For the diaphragm thickness measurements, the investigators used right hemidiaphragm with the linear transducer located between the anterior and middle axillary lines around the ninth intercostal space, in the diaphragmatic apposition zone (29,30). For the rectus abdominis thickness measurements the investigators used the linear transducer positioned 2 cm to the right and 2 cm above the umbilical scar. The external oblique, internal oblique and transverse muscles of the abdomen can be identified as three parallel layers, usually best visualized on the anterior axillary line, midway between the lower edge of the rib cage and the iliac crest (15,16) The window will be obtained in B-moded, and the measurement performed in M-mode. For the measurement of the thickening fraction, the investigators will use the formula ((Eins - Eex) /Ex) x 100), where Eins = thickness obtained at the end of inspiration and Eex = thickness obtained at the end of expiration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchiolitis
* Use of HFNC

Exclusion Criteria:

* Patients diagnosed with chronic diseases

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
diaphragm thickening fraction | during procedure
  to evaluate the diaphragm thickening fraction through ultrasound in infants with bronchiolitis using HFNC at 4 different flow rates, whether the diaphragm thickening fraction changes when the flow rate is changed
abdominal muscle thickening fraction | during procedure
  to evaluate the abdominal muscle thickening fraction through ultrasound in infants with bronchiolitis using HFNC at 4 different flow rates, whether the abdominal muscle thickening fraction changes when the flow rate is changed
EELZ (end-expiration lung impedance) | during procedure
  to evaluate the EELZ through electrical impedance tomography in infants with bronchiolitis using HFNC at 4 different flow rates, whether there is a change in the EELZ when the flow rate is changed

CONTACTS AND LOCATIONS:
Overall Officials: Milena S Nascimento, Principal Investigator — Hospital Israelita Albert Einstein; Celso M Rebello, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Eisntein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
This study will be in partnership with Childrens Hospital Los Angeles. The anonymized database will be shared containing all variables described in the methodology
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be shared after the inclusion of patients until the analysis of the results is completed
Access Criteria: All data will be compiled and managed in the electronic data capture system "Research Electronic Data Capture" (REDCap) hosted on the servers of Hospital Israelite Albert Einstein (HIAE) (33). All data, when made available to the project team, will be made available in a de-identified form in order to protect the participant's identity and guarantee the integrity of the data.